CLINICAL TRIAL: NCT03622840
Title: Impact of Individual Cognitive Remediation for Parkinson's Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Completed
Sponsor: New York Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: BHS-1379
Record Dates: First submitted 2018-06-20; First posted 2018-08-09 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Cognitive Impairment; Parkinson Disease
Keywords: Cognitive Remediation
MeSH Terms: conditions — Cognitive Dysfunction; Parkinson Disease | interventions — Cognitive Remediation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parkinson's disease patients with cognitive impairment (Other): Online cognitive remediation program.
  Interventions: Behavioral: Cognitive Remediation

INTERVENTIONS:
Behavioral: Cognitive Remediation — Weekly 30-45mins Cognitive Remediation Sessions over 11 weeks
  Other Names: Brain.HQ

SUMMARY:
This is an interventional clinical trial that will be conducted as a pilot project. Investigators hope to conduct the study to obtain at least 10 study completers.

The plan is to screen 20 Parkinson's Disease (PD) patients attending the Academic Health Care Center (AHCC) at NYIT College of Osteopathic Medicine clinic and enroll the eligible candidates based on the inclusion and exclusion criteria. Subjects will have 11 study visits over the 11-week period. Subjects cognition will be assessed using a paper-based Test of Memory and Learning (TOMAL) tool. The same tool will be used to asses and compare the cognition at baseline, and end study visits. The weekly 30-mins of cognitive remediation exercises will be done using the Brain. HQ cognitive remediation software.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be between 40 and 75 years old (including both ages) at the time of study screening.
2. Subjects must have a diagnosis of Parkinson's Disease by a physician.
3. Subjects must demonstrate adequate decisional capacity, in the judgment of the consenting study staff member, to make a choice about participating in this research study.
4. Subjects must have been clinically stable (non-acute) for 2 weeks prior to consent; in the judgment of the Investigator.
5. Subjects with a cognition level between Impaired and Average (scaled score between 4-12 or Index Score between 70-110) based on TOMAL Cognitive assessment at Visit 1
6. Subjects must have the visual, auditory, and motor capacity to use the intervention in the judgment of the Principal Investigator.

Exclusion Criteria:

1. Subjects who are participating in a concurrent research study or another interventional clinical trial 30 days prior to consenting.
2. Subjects having a history of mental retardation or pervasive developmental disorder; or other co-morbid neurological disorder (e.g., epilepsy.)
3. Subjects who appear to be intoxicated or under the influence of a controlled substance on any day of assessment must be rescheduled and may be discontinued based upon the discretion of the investigator
4. Subjects on medications that affect the cognition in the last 12 hours prior to the study visits that assess the cognitive functions

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Change of Test of Memory and Learning (TOMAL) score | Baseline and 11 weeks
  Paper based memory and attention test administered at the beginning and end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Anu Raj, Psy.D, Principal Investigator — New York Institute of Technology College of Osteopathic Medicine
Locations (1):
- New York Institute of Technology College of Osteopathic Medicine, Old Westbury, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided